CLINICAL TRIAL: NCT03678922
Title: The Danish Child and Adolescent Musculoskeletal Pain (ChiBPS) Cohort: Protocol for a Prospective Nationwide Cohort Study in General Practice
Acronym: ChiBPS
Status: Completed | Type: Observational
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Negar Pourbordbari, Doctor of medicine, Aalborg University
Other Study IDs: ChiBPS-Prot
Record Dates: First submitted 2018-09-04; First posted 2018-09-20 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Musculoskeletal Pain
Keywords: musculoskeletal pain; adolescents; children; prognosis; general practice; bio-psycho-social
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Musculoskeletal (MSK) pain in adolescents is much more persistent than commonly appreciated. It has previously been described as a self-limiting condition, but several studies indicate otherwise. In a cohort study of 564 11-year olds with weekly MSK pain, 50% of the participants still reported pain after one year. Prospective cohort studies of adults in general practice show that 16-32% of patients with knee pain still have pain after a year. In accordance with this, Kastelein et al. found that 21% of 12 to 35-year-old patients had knee pain six years after initial general practitioner (GP) contact. Collectively, these studies highlight that a significant proportion of adolescents will continue to report pain even years after the initial onset of pain.

Can the adolescents with a high risk of MSK pain at follow-up be investigated? Our recent systematic review on children and adolescents with MSK pain indicates that female sex, depression, anxiety, and parental pain are associated with a higher risk of MSK pain at follow-up. However, the validity of these prognostic factors may be questioned as they have been tested in single cohorts and not validated in new external cohorts. Moreover, in accordance with our results, other studies identify emotional problems, psychological symptoms, and frequent exercise associated to a higher risk of MSK pain at follow-up. Given the paucity of high-quality evidence for prognostic factors in childhood and adolescent MSK pain, robust studies are needed to further explore prognostic factors in this population. The investigators want to follow up on this need and conduct a cohort study with a similar aim as in their review; to investigate prognosis in youth MSK pain. In this cohort study, the investigators will limit their participant group to those who are 8-19 years old, because the participants have to be able to provide self-reported data on a questionnaire. Participants aged 0-7 years will not be included as they will have difficulties in doing so and because they i) only represent 2% of all patients consulting GPs in Denmark, with a musculoskeletal complaint and ii) were sparsely represented in our systematic review which included a total of 23.933 patients.

At present we lack age-specific prognostic factors in adolescents with MSK pain, although multiple prognostic factors have been identified in adult MSK pain. One systematic review found that higher pain severity upon presentation to the GP, longer pain duration, multiple-site pain, anxiety and/or depression, higher somatic perceptions and/or distress, low social support, higher baseline disability, and greater movement restriction were all associated with a poor prognosis. Systematic reviews on adult knee pain suggest an association between low/middle education level, non-skeletal comorbidity, duration of knee symptoms of > 3 months, bilateral knee symptoms, self-reported warm knee, history of non-traumatic knee symptoms, valgus alignment and an unfavorable prognosis. Similar to findings in patients with adult low back pain, there was high evidence that fear-avoidance beliefs and meagre social support at work were associated with an poor prognosis.

If future studies are to tailor and target treatment for the adolescents with the highest risk of long-standing MSK pain, there is a need to identify prognostic factors for an unfavorable prognosis. The aim of this prospective cohort study is to identify the most important prognostic factors for adolescents with MSK pain in general practice.

DETAILED DESCRIPTION:
This study is a prospective cohort study. Setting: Danish general practice clinics across Denmark. We have no interventions for this study. Patients will be followed from their initial pre-recruitment GP consultation and onwards. The pre-defined follow-up assessments are 3, 6 (primary), and 12 months, but the cohort will be followed continuously onwards every 1-5 years.

The aim is to recruit a sample that represents the Danish child and adolescent population with musculoskeletal pain.

The GP is suggested ways of recruitment, in order to choose which best suits the infrastructure of the individual clinic.

Recruitment by an employee:

The employee executes the recruitment process with a screen of all scheduled patients for that day. This prior to the first consultation of the day. The eligibility screening has two criteria: 1. Cause for consultation including a MSK pain complaint and 2. Age 8 to 19 years. The word MSK is written next to the names of all eligible patients to indicate and remind the employee or the consulting GP to hand out the questionnaire to the patient, before they leave the clinic.

Recruitment by the GP:

The GP screens the schedule for the day, and indicates eligibility with the word MSK written next to the patient name.

When consulting a patient with the indicated MSK, the GP is reminded to hand the patient the patient material. This can be done, prior, during or in the end of a consultation while the patient is getting dressed.

The patient hands in the completed questionnaire to an employee of the clinic, who stores it in a locked place. NP or her assistant will collect this in agreement with the clinic.

The child must first be included in the study in order for his/her parent(s) to be eligible. Of included children, data will be requested from parents during a time window of two weeks from the time of Part-Quest (participant questionnaire). The investigators are not selective as to if and how many of the parents wish to participate. Parents declining participation will not cause withdrawal of the childs' eligibility or inclusion.

Participants will be followed from their initial GP consultation initiating the inclusion and onwards. The pre-defined follow-up assessments are 3, 6 (primary), and 12 months, but the cohort will be followed continuously onwards every 1-5 years. At follow-up, a research assistant working together with and supervised by NP (Negar Pourbordbari) will contact the participants on phone, to remind them of the follow-up questionnaire they will receive by e-mail. A similar process will be repeated at all follow-up time points.

All included participants will be registered at eligibility screen, acquired written consent, and assessments, the latter collected at both baseline and follow-up time points.

With the primary outcome the investigators aim to capture pain that interferes with their everyday lives and collect the location of pain. The patient characteristics (exposures) are based on results from our systematic review, used in other studies (when including references).

The specific wording in the outcomes and throughout the questionnaire has been pilot tested among similar aged kids and adolescents.

The sample-size in this study was determined using the two following rationales: 1) a sample-size large enough to test and replicate the analyses from previous studies on. Given the prior odds (0.5, 1, 2) of follow-up MSK pain for patients, using estimates for the prognostic factors female sex, high disability index, multisite pain, and maximum HFAQ (Hannover Functional Ability Questionnaire) from our systematic review. The investigators gained an estimate of P-values according to sample size, for all factors individually (Appendix 8). Sample size of 500 patients, would result in an estimate of P-values below 0.05 for all prognostic factors and 2) investigate a range of new prognostic factors related to the sparsely investigated ethnicity and socioeconomic status. As no one has yet tested any of these potential important prognostic factors, and never in a general practice setting, the investigators decided on 500 subjects. The 500 subjects was decided based on 250 cases (50% will assume to continue to experience pain at our primary follow-up time) giving approximately 125 cases per prognostic factor (500/number of prognostic factors). The results from this analysis will be considered as explorative as no studies have previously been conducted in a general practice setting. Again, assuming 50% has pain at follow-up and 20 events for each to be tested factor are needed. The model should allow for 10-15 variables in a multivariable logistic regression analysis. This would lead to a sample size of 480. Assumed, 5% is lost to follow-up and we have a sample-size of 504 included participants. Given the high prevalence of MSK pain at follow-up, this sample-size is feasible to include.

The investigators use three questionnaires in data collection of patient and parent characteristics: participant baseline questionnaire (Part-Quest-base) (Appendix 2), participant follow-up questionnaire (Part-Quest-follow-up) (Appendix 3), and the parent questionnaire (Pare-Quest) (Appendix 4).

In relation to our previous study, all these factors have an interest as to whether they present as prognostic factors in MSK pain at follow-up.

The questionnaires will be pilot tested among target participants; Part-Quest among 8-19-year-olds with MSK pain and the Pare-Quest among parents to children with MSK pain.

Our questionnaires wil be cross-cultural adaptive for participants with poor Danish language skills, insufficient to comprehend the original Danish questionnaires. In the process of translation and validation, we will translate our questionnaires both linguistically and culturally. Our three questionnaires and our bulletin will be translated from English to Danish, which is the mother tongue of the majority of our prospective participants.

The questionnaires, will be handed to the participants and their parents in paper. If they are not able to complete the questionaires while still in the clinical setting (waiting room) and hand them to the secretary when completed, they may at a later point in time (no later than seven days) hand them in at the clinic. Seven days of response time, will be applicable also for follow-up questionnaires, before a reminder is sent out. In contrary to the baseline questionnaire, the follow-up questionnaires will be administered to the participants and parents through e-mail. If for some reason a participant do not respond within the given time limit, he/she will be reminded by e-mail or phone. This will be executed by the assistant, to ensure a satisfactory follow-up rate.

Retrieved data from both baseline and follow-up participant questionnaires and parent questionnaire will be handled according to the Danish Data Protection Agency.

Descriptive results will be stratified by sex and MSK pain type, presented with their central estimate and appropriate measure of dispersion (95% confidence interval CI). All descriptive statistics and test will be reported in accordance to the recommendations of the STROBE statement.

We will test the univariate association between each potential prognostic factor as well as combining the factors in a multivariable model to show the individual contributions.

The primary analysis will be done on those who has a first time consultation with their GP concerning their current MSK pain, but all consultations will be included.

The full statistical analysis plan will be developed concurrently and will be finalized before the last patient is enrolled. Information bias will be minimised by use of identical questionnaires for all patients included, e.g. by asking both Danes and non-Danes whether they feel Danish or not.

The adolescents included in the ChiBPS cohort will receive usual care, i.e. as usually administered at their GP. This study will not intervene in the diagnostic and therapeutic process.

Since our target audience is general practitioners, our prognostic factors must be applicable in a GP setting in relation to the terminology they are presented in as results of this study. In order to gain recognition of this, NP will create a temporary subgrouping, based on the prognostic factors from our recent systematic review. She will convey this subgrouping to a focus group consisting of 15 clinically experienced, Danish GP physician peers for feedback on the suggested terminology in subgrouping of the prognostic factors. She will ask for any concerns in comprehension including any suggestions towards an easy digestible language, in the context of general practice.

ELIGIBILITY:
Inclusion Criteria:

* 8 to 19 years
* Self-reported musculoskeletal pain Traumatic pain caused by soft tissue damage, contusion or otherwise (excluding fracture), will be included.

Exclusion Criteria:

* 0-7 or 20+ years
* Self-reported musculoskeletal pain due to tumor, fracture, infection, or systemic and neurological causes.

Parental participation will only be eligible after inclusion of their child. If a child is not eligible, or parental consent is not acquired on behalf of the child or adolescent <15 years of age, the parent will not be eligible for inclusion.

Ages: 8 Years to 19 Years | Sex: All
Age Groups: Child, Adult
Study Population: The children and adolescents must have self-reported MSK pain at the time of recruitment and consult the GP in relation to their MSK pain. The primary reason for consultation may not necessarily be listed as MSK pain, but to be eligible for inclusion, MSK pain must be mentioned during the consultation with the GP. We do not have a pre-defined minimum or maximum MSK pain duration as a eligibility criteria and patients are eligible whether or not they have previously consulted their GP for their current MSK complaint.
  We define MSK pain according to the International Association for the Study of Pain (IASP) as: "pain arisen from muscle, tendon, bone, and joint". Pain due to tumor, fracture, infection, or systemic and neurological cause will be excluded. Types of pain will be labelled according to the region affected, e.g. back pain, neck pain, shoulder pain, knee pain etc
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Activity limiting pain | 6 months
  Have you experienced pain in the past two weeks that have lead you to not being able to participate in play in the school yard or sparetime activities (ex. football or other sparetime activity? yes/no
Location of activity limiting pain (must include same location as baseline) | 6 months
  If yes to Primary Outcome 1: Please mark the areas of your body where you have had pain during the past two weeks (pictured a mannequin)

SECONDARY OUTCOMES:
Pain intensity depicted on a NRS (11 point numeric rating scale) | 6 months
  Pain intensity depicted on a NRS (11 point numeric rating scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Aalborg, Denmark

REFERENCES:
- [Derived] Pourbordbari N, Jensen MB, Olesen JL, Holden S, Rathleff MS. Prognosis and bio-psycho-social prognostic factors in children and adolescents with musculoskeletal pain consulting general practice. Eur J Pediatr. 2025 Jun 2;184(6):384. doi: 10.1007/s00431-025-06217-2. PMID 40455265
- [Derived] Pourbordbari N, Jensen MB, Olesen JL, Holden S, Rathleff MS. Bio-psycho-social characteristics and impact of musculoskeletal pain in one hundred children and adolescents consulting general practice. BMC Prim Care. 2022 Jan 25;23(1):20. doi: 10.1186/s12875-022-01628-8. PMID 35172756

DOCUMENTS (1):
  • Study Protocol (2018-08-20): https://cdn.clinicaltrials.gov/large-docs/22/NCT03678922/Prot_000.pdf